CLINICAL TRIAL: NCT01453465
Title: Gene Expression (GE) and MicroRNA (MIRNA) Expression Profiles of Malignant Rhabdoid Tumors (MRT) of the Kidney (RTK) and Atypical Teratoid Rhabdoid Tumor (ATRT)
Brief Title: Biomarker Study in Samples From Patients With Malignant Rhabdoid Tumor of the Kidney or Atypical Teratoid Rhabdoid Tumor
Status: Withdrawn | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: ABTR12B1; NCI-2011-03468 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000712872; ABTR12B1; COG-ABTR12B1; ABTR12B1 (Other: Childrens Oncology Group); ABTR12B1 (Other: CTEP)
Record Dates: First submitted 2011-10-01; First posted 2011-10-17 (Estimated); Last update posted 2018-08-07 (Actual); Status verified 2017-10

CONDITIONS: Childhood Atypical Teratoid/Rhabdoid Tumor; Rhabdoid Tumor of the Kidney
MeSH Terms: conditions — Rhabdoid Tumor

GROUPS / COHORTS (1):
- Ancillary-Correlative (gene expression profile, miRNA profile): Archived tumor tissue samples are analyzed for gene expression profile and microRNA profile.
  Interventions: Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This research trial studies biomarkers in samples from patients with rhabdoid tumor of the kidney and atypical teratoid rhabdoid tumor. Studying biomarkers of tissue samples from patients with cancer in the laboratory may help doctors learn more about changes the occur in DNA and identify biomarkers related to cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if there are molecular differences between rhabdoid tumor of the kidney (RTK) and the atypical teratoid rhabdoid tumor (ATRT).

OUTLINE:

Archived tumor tissue samples are analyzed for gene expression profile and microRNA profile.

ELIGIBILITY:
Inclusion Criteria:

* Samples of RTK and ATRT provided by the Children?s Oncology Group (COG)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-11-01 (Actual); Primary Completion 2011-12-01 (Actual)

PRIMARY OUTCOMES:
Molecular differences between RTK and the ATRT | Up to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Simone Sredni, Principal Investigator — Children's Oncology Group
Locations (1):
- Childrens Oncology Group, Philadelphia, Pennsylvania, United States